CLINICAL TRIAL: NCT01358773
Title: Multiprofessional Impact on Body Composition, Central and Peripheric Adiposity, Lipid Profile, Hormonal Regulation, Lung, Sleep and Humor Disorders in Adolescents
Brief Title: The Effect of 1 Year of Multiprofessional Therapy on Obesity
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ana R. Damaso (Other)
Collaborators: Raquel Munhoz da Silveira Campos (Unknown); Sofia Emanuelle Castro (Unknown); Ana Claudia Pelissari Kravchychyn (Unknown)
Responsible Party: Sponsor-Investigator, Ana R. Damaso, Associated Professor, Federal University of São Paulo
Organization: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #0135/04
Record Dates: First submitted 2010-12-03; First posted 2011-05-24 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Obesity
Keywords: Obesity; Therapy; Interdisciplinary
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle counseling (Other): Obese adolescents are encouraged to improve their lifestyle
  Interventions: Other: multidisciplinary intervention

INTERVENTIONS:
Other: multidisciplinary intervention — Comparison of the polysomnography results, blood collection parameters, resting metabolic rate values, body composition variables, carotid artery thickness values, abdominal and subcutaneous fat and lung function variables baseline, middle and at the end of the one year of interdisciplinary weight loss program combined exercise training with physiotherapy, clinical, nutritional and psychological therapies.
  Other Names: Interdisciplinary therapy

SUMMARY:
Obese adolescents are submitted to a multiprofessional weight loss program, which is formed by doctors, nutritionists, physiotherapists, psychologists,and physiologists. The volunteers have intervention 3 times a week during one year, where they practice exercises, have nutrition and psychology counseling, and physiotherapy orientation. Once a month they have an appointment with the doctor. The hypothesis of this study is that a multiprofessional therapy is able to improve anthropometric and biochemical parameters, and also the quality of life of obese adolescents.

DETAILED DESCRIPTION:
The volunteers are submitted to 10 exams (electrocardiogram, polysomnography, blood collection, body composition, rest metabolic rate, DXA, abdominal and carotid ultrasonography, lung function evaluation, ergospirometric test) 3 times a year (baseline, middle and at the end of the year). They also answer nutrition, sleep and psychology questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* present obesity ( BMI > 95th)
* aged between 15-19 years old
* be able to practice exercise

Exclusion Criteria:

* pregnancy
* use of drugs
* secondary obesity

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2004-02; Primary Completion 2004-12 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Body composition | six months
  The body composition was measured by plethysmography and by densitometry.

SECONDARY OUTCOMES:
visceral and subcutaneous fat were analyzed by ultrasound | six months
  The visceral and subcutaneous fat were analyzed by ultrasound
Serum analysis | six months
  The serum analysis was done by blood samples that were collected at the outpatient clinic around 8 a.m. after an overnight fast by a skilled and qualified technician.
Lung function | six months
  The lung function was measured with a spirometer EasyOne® model 2001 (Zurich, CH) according to American Thoracic Society criteria.
Arterial intima-media thickness | six months
  The arterial intima-media thickness was measured by High-resolution ultrasound equipment with a 7-14 MHz linear array transducer.
Sleep parameters | six months
  The sleep parameters were evaluated by polysomnography and specific questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Ana R Dâmaso, PhD, Principal Investigator — Universidade Federal de São Paulo- UNIFESP - Escola Paulista de Medicina - EPM
Locations (1):
- CEPE, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Roche J, Corgosinho FC, Damaso AR, Isacco L, Miguet M, Fillon A, Guyon A, Moreira GA, Pradella-Hallinan M, Tufik S, Tulio de Mello M, Gillet V, Pereira B, Duclos M, Boirie Y, Masurier J, Franco P, Thivel D, Mougin F. Sleep-disordered breathing in adolescents with obesity: When does it start to affect cardiometabolic health? Nutr Metab Cardiovasc Dis. 2020 Apr 12;30(4):683-693. doi: 10.1016/j.numecd.2019.12.003. Epub 2019 Dec 16. PMID 32008915
- [Derived] Masquio DC, de Piano A, Campos RM, Sanches PL, Carnier J, Corgosinho FC, Netto BD, Carvalho-Ferreira JP, Oyama LM, Oller do Nascimento CM, Tock L, de Mello MT, Tufik S, Damaso AR. Reduction in saturated fat intake improves cardiovascular risks in obese adolescents during interdisciplinary therapy. Int J Clin Pract. 2015 May;69(5):560-70. doi: 10.1111/ijcp.12573. Epub 2014 Oct 9. PMID 25296762
- [Derived] Grotti Clemente AP, Molin Netto BD, Ganen Ad, Tock L, Arisa Caranti D, de Mello MT, Tufik S, Damaso AR. Cut-Off Values of Visceral Adiposity to Predict NAFLD in Brazilian Obese Adolescents. J Nutr Metab. 2013;2013:724781. doi: 10.1155/2013/724781. Epub 2013 Dec 7. PMID 24381750
- [Derived] de Piano A, de Mello MT, Sanches Pde L, da Silva PL, Campos RM, Carnier J, Corgosinho F, Foschini D, Masquio DL, Tock L, Oyama LM, do Nascimento CM, Tufik S, Damaso AR. Long-term effects of aerobic plus resistance training on the adipokines and neuropeptides in nonalcoholic fatty liver disease obese adolescents. Eur J Gastroenterol Hepatol. 2012 Nov;24(11):1313-24. doi: 10.1097/MEG.0b013e32835793ac. PMID 22932160
- [Derived] Corgosinho FC, de Piano A, Sanches PL, Campos RM, Silva PL, Carnier J, Oyama LM, Tock L, Tufik S, de Mello MT, Damaso AR. The role of PAI-1 and adiponectin on the inflammatory state and energy balance in obese adolescents with metabolic syndrome. Inflammation. 2012 Jun;35(3):944-51. doi: 10.1007/s10753-011-9397-2. PMID 22038064